CLINICAL TRIAL: NCT04244266
Title: Observational Study of the Pharmacological Reversal of the Residual Neuromuscular Blockade in Bariatric Surgery
Brief Title: Observational Study in Bariatric Surgery
Acronym: NEOCURE
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NEOCURE; 2019-A02647-50 (Other: IDB-RCB)
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Obesity; Neostigmine; Residual Neuromuscular Blockade
MeSH Terms: conditions — Obesity; Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Ideal Body Weight: groups of patients divided according to neostigmine dose weight, ideal body weight (IBW)
  Interventions: Other: NO INTERVENTION, it is an observational study
- Total Body Weight: groups of patients divided according to neostigmine dose weight, total body weight (TBW),
  Interventions: Other: NO INTERVENTION, it is an observational study
- Adjusted Body Weight: groups of patients divided according to neostigmine dose weight, , adjusted body weight (ABW)
  Interventions: Other: NO INTERVENTION, it is an observational study

INTERVENTIONS:
Other: NO INTERVENTION, it is an observational study — No intervention

SUMMARY:
Obesity in the world represents a growing share of the general population. At hospital, the management of these patients could be problematic especially when calculating the drug dosage.

According to the French guidelines, neostigmine, a cholinesterase inhibitor, should be used to reverse a residual neuromuscular blockade at a dose of 0.4 mg/kg of total body weight in non-obese patients. In morbidly-obese patients, with the modification of the fat/lean mass ratio, the optimal dose of neostigmine is non-consensual. To calculate the dose of neostigmine, some anesthesiologists use the total body weight, others use the ideal body weight and others use the adjusted body weight.

Due to this practice variability, It may be useful to observe the mean time to recovery of neuromuscular blockade and side effects after pharmacological reversal according to the dosage of neostigmine.

ELIGIBILITY:
Inclusion Criteria*:

* Adult obese patients (≥ 18 years and BMI ≥ 35 Kg/m²), both sexes
* Any elective bariatric surgery
* Neuromuscular blockade with rocuronium
* Maintenance of anesthesia with a halogenated agent
* Free patient, without guardianship or subordination
* Patients with a social security coverage
* No opposition given by the patient after clear and fair information

Exclusion Criteria*:

* Patients with hypersensitivity to the active substance or to other derivatives, or to any of the excipients of neostigmine,
* Emergency surgery,
* Severe renal and / or hepatic insufficiency,
* Persons benefiting from enhanced protection, namely pregnant women, breastfeeding women, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection and finally sick people in emergency situation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients whose BMI will be higher than 35 kg/m²
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Compare the mean delay to recovery of neuromuscular blockade after pharmacological reversal according to the dosage of neostigmine administered to the patient (on TBW, IBW or ABW | Few minutes after injection of neostigmine
  Delay between the injection of neostigmine T0 and obtain a ratio between the 4th and the 1st response (T4/T1) by "Four-Train Stimulator" (TOF) ≥ 0.9

SECONDARY OUTCOMES:
Compare the frequence of side effects according to the dosage of neostigmine administered (on TBW, IBW or ABW) | Within one hour after the injection of neostigmine
  Occurrence of bradycardia defined by a heart rate <50 beats per minute in the hour following the injection of neostigmine Occurrence of bronchospasm defined by a desaturation over 92% and sibilants to the auscultation within one hour after neostigmine injection.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No